CLINICAL TRIAL: NCT01305096
Title: Effects of Yoga on Objective and Self-reported Health Indicators Among Female and Male Individuals
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: Region Stockholm (Other Government); Stockholm University (Other)
Responsible Party: Principal Investigator, Per Wandell, Professor, Karolinska Institutet
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 2011/248-31/1
Record Dates: First submitted 2011-02-25; First posted 2011-02-28 (Estimated); Last update posted 2014-10-24 (Estimated); Status verified 2014-10

CONDITIONS: Stress, Psychological, Physiological
Keywords: heart rate variability; oxygen uptake; heart rate recovery; perceived stress; sleep; blood pressure; body mass index; body weight; hand grip strength; sleep quality; subjective health complaints; blood lipids; salivary cortisol; blood sugar; HbA1C; Adiponectin; Leptin; Adipolipoproteins; blood proteins; cytokines; insomnia; sleeplessness; yoga
MeSH Terms: conditions — Body Weight; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Yoga group (Experimental): Participants in this group will take part in six to eight weeks of yoga classes. The classes will be held once a week and each class will be approximately one hour long. The classes will consist of yoga inversions, sun salutations and other yoga postures with deep breathing.
  Interventions: Other: Yoga intervention
- Control group (No Intervention): Matched control

INTERVENTIONS:
Other: Yoga intervention — 6 weeks of yoga postures, once a week for 60 minutes in a group session with a yoga teacher.
  Arms: Yoga group

SUMMARY:
The purpose of this study is to determine whether inversions (specific yoga postures in which the heart is higher than the head) and other dynamic and static yoga postures affect heart rate variability, oxygen uptake, blood pressure, blood parameters and other objective measures of health, and a variety of subjective and objective measures of health in female and male individuals in Sweden.

DETAILED DESCRIPTION:
This randomized, controlled trial involving 44 male and females in Sweden will investigate whether yoga inversions and semi-inversions and other dynamic and static yoga postures will affect the following variables: heart rate variability, oxygen uptake, anthropometric variables, common symptoms in general practice, sleepiness, sleep quality and recovery/recuperation after sleep, blood pressure, blood lipids, blood proteins, blood sugar, salivary cortisol, hand grip strength, relaxation and recovery perceived stress, self-rated health, rating of perceived exertion, satisfaction with life, and work-family conflict.

Participants will be divided into an intervention group and a passive control group. The intervention group will participate in six to ten weeks of yoga classes. The classes will be held 1-2 times a week for approximately one hour each and will include yoga poses and breathing techniques. The control group will not participate in any intervention but will conduct their lives as usual.

The variables will be assessed at baseline; at the end of the intervention; and three, six, and twelve months after the end of the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Aged 20-40 years old

Exclusion Criteria:

* Aged 40 or more years
* Takes medication for high blood pressure or other strong medication
* Recently had an operation
* Diagnosed with eye disease (e.g., glaucoma)
* Diagnosed with depression or burnout syndrome
* Diagnosed with serious back or neck problems
* Participates in intense physical activity more than once a week
* Has digestive problems such as acid reflux
* Serious disorder that affects the ability to do the yoga postures

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2011-03; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Change in heart rate variability | Baseline and at the end of the 8-week intervention
  We will measure the change in this variable over time. The first measurement will be at baseline and the second at the end of the 8-week intervention (main measurement). If and only if there are effects after the 8-week intervention, we will follow up the participants at various intervals to determine how long the effects are sustained. These follow-ups will be conducted 3 months, 6 months, and 12 months after the end of the intervention.
Change in oxygen uptake | Baseline and at the end of the 8 week intervention
  We will measure the change in this variable over time. The first measurement will be at baseline and the second at the end of the 8-week intervention (main measurement). If and only if there are effects after the 8-week intervention, we will follow up the participants at various intervals to determine how long the effects are sustained. These follow-ups will be conducted 3 months, 6 months, and 12 months after the end of the intervention.

SECONDARY OUTCOMES:
Change in anthropometric variables | Baseline and at the end of the 8-week intervention
  Anthropometric variables include height, weight, waist-to-hip ratio, and body mass index(BMI). We will measure the change in these variables over time. The first measurement will be at baseline and the second at the end of the 8-week intervention (main measurement). If and only if there are effects after the 8-week intervention, we will follow up the participants at various intervals to determine how long the effects are sustained. These follow-ups will be conducted 3 months, 6 months, and 12 months after the end of the intervention.
Change in common symptoms in general practice | Baseline and at the end of the 8-week intervention
  We will use the Common Symptoms in General Practice Index to measure how often over the past four weeks participants have experienced the fifteen most common health-related symptoms and complaints. The first measurement will be at baseline and the second at the end of the 8-week intervention (main measurement). If and only if there are effects after the 8-week intervention, we will follow up the participants at various intervals to determine how long the effects are sustained. These follow-ups will be conducted 3 months, 6 months, and 12 months after the end of the intervention.
Change in level of sleepiness and measures of recovery or recuperation after sleep | Baseline and at the end of the 8-week intervention
  The Karolinska Sleepiness Scale will be used to measure this outcome variable. This scale measures degree of wakefulness at bedtime and after waking in the morning. The first measurement will be at baseline and the second at the end of the 8-week intervention (main measurement). If and only if there are effects after the 8-week intervention, we will follow up the participants at various intervals to determine how long the effects are sustained. These follow-ups will be conducted 3 months, 6 months, and 12 months after the end of the intervention.
Change in blood pressure | Baseline and at the end of the 8-week intervention
  We will measure the change in this variable over time. The first measurement will be at baseline and the second at the end of the 8-week intervention (main measurement). If and only if there are effects at the end of the 8-week intervention, we will follow up the participants at various intervals to determine how long the effects are sustained. These follow-ups will be conducted 3 months, 6 months, and 12 months after the end of the intervention.
Change in hand grip strength | Baseline and at the end of the 8-week intervention
  We will measure the change in this variable over time. The first measurement will be at baseline and the second at the end of the 8-week intervention (main measurement). If and only if there are effects after the 8-week intervention, we will follow up the participants at various intervals to determine how long the effects are sustained. These follow-ups will be conducted 3 months, 6 months, and 12 months after the end of the intervention.
Change in measures of relaxation and recovery | Baseline and at the end of the 8-week intervention
  We will measure the change in these variables over time. The first measurement will be at baseline and the second at the end of the 8-week intervention (main measurement). If and only if there are effects after the 8-week intervention, we will follow up the participants at various intervals to determine how long the effects are sustained. These follow-ups will be conducted 3 months, 6 months, and 12 months after the end of the intervention.
Change in perceived stress | Baseline and at the end of the 8-week intervention
  The Perceived Stress Scale will be used to measure this variable. The first measurement will be at baseline and the second at the end of the 8-week intervention (main measurement). If and only if there are effects after the 8-week intervention, we will follow up the participants at various intervals to determine how long the effects are sustained. These follow-ups will be conducted 3 months, 6 months, and 12 months after the end of the intervention.
Change in self-rated health | Baseline and at the end of the 8-week intervention
  We will measure the change in this variable over time. The first measurement will be at baseline and the second at the end of the 8-week intervention (main measurement). If and only if there are effects after the 8-week intervention, we will follow up the participants at various intervals to determine how long the effects are sustained. These follow-ups will be conducted 3 months, 6 months, and 12 months after the end of the intervention.
Change in rating of perceived exertion | Baseline and at the end of the 8-week intervention
  We will measure the change in this variable over time. The first measurement will be at baseline and the second at the end of the 8-week intervention (main measurement). If and only if there are effects after the 8-week intervention, we will follow up the participants at various intervals to determine how long the effects are sustained. These follow-ups will be conducted 3 months, 6 months, and 12 months after the end of the intervention.
Change in satisfaction with life | Baseline and at the end of the 8-week intervention
  This variable will be measured with the Satisfaction With Life Scale. The first measurement will be at baseline and the second at the end of the 8-week intervention (main measurement). If and only if there are effects after the 8-week intervention, we will follow up the participants at various intervals to determine how long the effects are sustained. These follow-ups will be conducted 3 months, 6 months, and 12 months after the end of the intervention.
Change in level of work-family conflict | Baseline and at the end of the 8-week intervention
  This variable will be measured with the Work-Family Conflict Scale. The first measurement will be at baseline and the second at the end of the 8-week intervention (main measurement). If and only if there are effects after the 8-week intervention, we will follow up the participants at various intervals to determine how long the effects are sustained. These follow-ups will be conducted 3 months, 6 months, and 12 months after the end of the intervention.
Change in HbA1C | Baseline and at the end of the 8-week intervention
  We will measure the change in this variable over time. The first measurement will be at baseline and the second at the end of the 8-week intervention (main measurement). If and only if there are effects after the 8-week intervention, we will follow up the participants at various intervals to determine how long the effects are sustained. These follow-ups will be conducted 3 months, 6 months, and 12 months after the end of the intervention.
Change in Apolipoproteins | Baseline and after the 8-week intervention
  We will measure the change in this variable over time. The first measurement will be at baseline and the second at the end of the 8-week intervention (main measurement). If and only if there are effects after the 8-week intervention, we will follow up the participants at various intervals to determine how long the effects are sustained. These follow-ups will be conducted 3 months, 6 months, and 12 months after the end of the intervention.
Change in Adiponectin/Leptin ratio | Baseline and at the end of the 8-week intervention
  We will measure the change in this variable over time. The first measurement will be at baseline and the second at the end of the 8-week intervention (main measurement). If and only if there are effects after the 8-week intervention, we will follow up the participants at various intervals to determine how long the effects are sustained. These follow-ups will be conducted 3 months, 6 months, and 12 months after the end of the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Per Wändell, MD, PhD, Professor, Study Chair — Karolinska Institutet; Petra Lindfors, PhD, Professor, Study Chair — Stockholm University; Malin Nygren, PhD, Study Chair — Karolinska Institutet; Lennart Gullstrand, PhD, Study Chair — Riksidrottsförbundet
Locations (1):
- Karolinska Institute, Stockholm, Sweden

REFERENCES:
- [Derived] Papp ME, Nygren-Bonnier M, Gullstrand L, Wandell PE, Lindfors P. A randomized controlled pilot study of the effects of 6-week high intensity hatha yoga protocol on health-related outcomes among students. J Bodyw Mov Ther. 2019 Oct;23(4):766-772. doi: 10.1016/j.jbmt.2019.05.013. Epub 2019 May 15. PMID 31733760